CLINICAL TRIAL: NCT00721487
Title: A Case Series of Investigator-Identified Fluconazole Failures: Outcome Characterization of Patients Who Fail to Respond to Fluconazole Treatment of Severe Infections Caused by Candida Albicans
Brief Title: Outcomes of Patients Who Fail to Respond to Fluconazole Treatment of Severe Candida Albicans Infections
Status: Completed | Type: Observational
Sponsor: CPL Associates (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Jerome Schentag, CEO, CPL Associates
Other Study IDs: MYCA-8F16
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Fungal Infection by Site
Keywords: C. albicans; fluconazole
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fluconazole: 30 evaluable patients hospitalized with severe infection caused by C. albicans, documented by standard clinical signs, symptoms, and radiology, and having failed at least four days of fluconazole therapy.
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Fluconazole — Patients hospitalized with severe infection caused by C. albicans, documented by standard clinical signs, symptoms, and radiology, and having failed at least four days of fluconazole therapy

SUMMARY:
The primary aims of this study are to identify and characterize the immediate consequences of patients who fail fluconazole treatment during the treatment of severe infection, and to determine if fluconazole failures are more frequently associated with fluconazole-resistant or fluconazole-susceptible strains of C. albicans.

DETAILED DESCRIPTION:
The primary aims of this study are to identify and characterize the immediate consequences of patients who fail fluconazole treatment during the treatment of severe infection, and to determine if fluconazole failures are more frequently associated with fluconazole-resistant or fluconazole-susceptible strains of C. albicans (i.e. does in vitro resistance matter?). Perhaps the breakpoints are not correct and need to be changed, as has recently happened with vancomycin.

A third objective is to calculate fluconazole PK/PD parameters such as AUIC, and compare the calculated AUIC values of patients who fail with fluconazole-susceptible vs fluconazole-resistant isolates. Specifically for fluconazole, the question here is whether dose matters, and can aggressive dosing offset higher MICs. Thus in all cases, we will also determine the AUIC of fluconazole in order to fully characterize the impact of dose chosen on the outcomes of treated patients who fail to respond to fluconazole. The clinical, microbiological, and pharmacoeconomic outcomes of patients who fail fluconazole therapy and are subsequently hospitalized with severe infections caused by C. albicans will be documented and described.

ELIGIBILITY:
Inclusion Criteria:

1. Medical history, clinical signs and symptoms, and radiological findings consistent with severe C. albicans infection. For example, the criteria for pneumonia are as follows:

   1. A core body temperature >38C [100.4F] or <36.1 C [97oF] or leukocytosis (blood leukocyte count >10,000 cells/mm3) or bandemia (>10% bands).
   2. Chest radiographic examination that shows a new or progressive infiltrate, consolidation, cavitation, or pleural effusion.
   3. Rales, dullness to percussion, or decreased breath sounds on physical examination of the chest, new onset of purulent sputum, or change in character of sputum.
2. A positive culture must demonstrate the presence of C. albicans, isolated from a properly obtained respiratory or blood sample, collected within 72 hours of admission to a hospital. All patients with respiratory cultures must produce sputum with Gram stain analysis indicating the relative absence of contaminating oropharyngeal squamous cells and the presence of a significant number of WBCs and morphologically distinct bacteria. Fluconazole sensitivity testing results must be available for the initial C. albicans isolate.
3. Must have received, and failed to respond to, at least 4 days of treatment with fluconazole.

4. Admitted to a hospital or ICU for treatment of a severe infection.

Exclusion Criteria:

1. Pregnant or lactating women
2. Cystic fibrosis
3. Life expectancy <3 months from underlying disease
4. Underlying lung carcinoma

Ages: 4 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a multi-center study of adult and pediatric patients hospitalized with severe infection caused by C. albicans. An announcement of this case series collection study will be sent to our ongoing list of primary care practitioners, hospitalists, specialists in infectious diseases, pulmonologists, clinical pharmacists, and other investigators throughout the USA.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Schentag, Pharm.D., Principal Investigator — CPL Associates, LLC; Joseph Paladino, Pharm.D., Principal Investigator — CPL Associates, LLC
Locations (1):
- CPL Associates,LLC, Buffalo, New York, United States